CLINICAL TRIAL: NCT00212342
Title: Phase 3,Placebo Controlled,Randomized,Double-Blinded,NSAID-Add-on,Clinical Trial of Mono-phase Low Dose Oral Contraceptive Pill for Treatment of Dysmenorrhea Associated With Endometriosis.
Brief Title: Efficacy and Safety Study of Low Dose Oral Contraceptive Pill to Treat Dysmenorrhea
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Nobelpharma (Industry)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: IKH-01-4
Record Dates: First submitted 2005-09-13; First posted 2005-09-21 (Estimated); Last update posted 2010-09-08 (Estimated); Status verified 2010-09

CONDITIONS: Dysmenorrhea
MeSH Terms: conditions — Dysmenorrhea | interventions — Norethindrone; Ethinyl Estradiol; Sugars

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor

ARMS (2):
- Norethisterone,Ethinylestradiol (Experimental)
  Interventions: Drug: Norethisterone,Ethinylestradiol
- Sugar pill (Placebo Comparator)
  Interventions: Drug: Sugar pill

INTERVENTIONS:
Drug: Norethisterone,Ethinylestradiol
  Arms: Norethisterone,Ethinylestradiol
Drug: Sugar pill
  Arms: Sugar pill

SUMMARY:
The purpose of this study is to determine whether combination oral contraceptive pill of Norethindrone & Ethinyl estradiol is effective in the treatment of dysmenorrhea associated with endometriosis.

ELIGIBILITY:
Inclusion Criteria:

* dysmenorrhea associated with endometriosis

Exclusion Criteria:

* severe hepatopathy
* pregnant woman

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2004-12; Primary Completion 2006-01 (Actual); Study Completion 2006-03 (Actual)

PRIMARY OUTCOMES:
patient response to treatment for dysmenorrhea associated with endometriosis,as evaluated by VRS

SECONDARY OUTCOMES:
changes in the VAS of dysmenorrhea.
changes in the VRS of non-menstrual pain.
changes in the VAS of non-menstrual pain.
changes in the clinical evaluation of pelvic induration.
changes in the size of ovarian endometrioma.

CONTACTS AND LOCATIONS:
Overall Officials: Naoki Terakawa, M.D.,Ph.D., Study Director — Tottori University,Tottori,Japan